CLINICAL TRIAL: NCT03094936
Title: Randomized Clinical Trial for Weight Regain Post-RYGB:Argon Plasma Coagulation Versus Argon Plasma Coagulation Plus Endoscopic Suture Technique
Brief Title: Clinical Trial for Weight Regain Post-RYGB: APC Versus APC Plus Endoscopic Suture Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Eduardo Guimarães Hourneaux de Moura, Director, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43405415000000068
Record Dates: First submitted 2015-09-03; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Other): This group own twenty patients who met all the inclusion criteria. These will be treated with APC.
  Interventions: Procedure: APC
- Group B (Active Comparator): This group own twenty patients who met all the inclusion criteria. These will be treated with APC plus Endoscopic Suture Technique (OverStitch TM).
  Interventions: Procedure: APC; Device: Endoscopic Suture Technique (OverStitch TM)

INTERVENTIONS:
Procedure: APC — Ablation of the dilated gastro-jejunal anastomosis with Argon Plasma Coagulation. This procedure induces cicatrization process around the stoma and propitiates its reduction.
Device: Endoscopic Suture Technique (OverStitch TM) — OverStitchTM Endoscopic Suturing System. Stitches will be placed per-orally with the aforementioned device around the dilated stoma in order to reduce the diameter of the anastomosis. In this group, ablation with APC will be done immediately before suturing.
  Other Names: Apollo Overstitch
  Arms: Group B

SUMMARY:
Obesity is a worldwide health and sociopolitical problem. Excessive body-weight currently affects over 50% of the Brazilian population. It has been well established that obesity is an independent health risk. Obese individuals are at increased to extremely high risk for many diseases and for early death relative to those with normal weights and waist circumferences. The increased disease susceptibility for this subset of patients includes hypertension, stroke, hyperlipidemia, sleep apnea, Type 2 diabetes, neoplasms, Gastro-Esophageal Reflux Disease, and musculoskeletal disorders.

Bariatric surgery is the most effective treatment for obesity. As bariatrics grow, the number of patients suffering from surgical-related complications also grows. One of the most worrisome long-term complications is weight regain, once the patient may be again affected by overweight-related comorbidities and face again pre-operative esthetic issues.

This trial focus on testing efficacy and safety of two endoscopic revisional procedures in patients suffering from weight regain following Roux-en-Y Gastric Bypass: Ablation with Argon Plasma Coagulation (APC) versus APC plus Endoscopic Full-thickness Suture (with Apollo Overstitch device). Pouch volume, gastric emptying and gut hormones changes will also be assessed.

DETAILED DESCRIPTION:
Obesity is a worldwide health and sociopolitical issue. Excessive body-weight currently affects over 50% of the Brazilian population and around 13% of all world population. It has been well established that obesity is an independent risk factor. Obese individuals are at increased risk of diseases and earlier death compared to those with normal weight and waist circumferences. The increased disease susceptibility of this subset of patients includes hypertension, stroke, hyperlipidemia, sleep apnea, Type 2 diabetes, neoplasms, GERD, and musculoskeletal disorders.

Obese patients and their physicians have increasingly turned to surgery to solve the excess weight issue and the frequent co-morbid conditions that impact their health and quality of life. Roux-en-Y Gastric Bypass (RYGB) and Laparoscopic Gastric Banding (LGB) comprise around 70% of all weight loss procedures performed every year. They induce significant and perennial weight loss and reduce or eliminate associated co-morbid diseases, including Type 2 diabetes. Despite improvements in postoperative morbidity and mortality rates over the years, (in part due to the use of a laparoscopic approach), these procedures still carry significant risk. Recent studies have shown mortality rates with RYGB as high as 1.9%, and complications associated with LGB as high as 13%. Nonetheless, a secondary bariatric procedure due to weight regain carries significant complication rates and worse outcomes, compared to the primary procedure. Consequently, less invasive techniques are needed to reduce such risks.

Gastric restriction is an important principle of both RYGB and LGB. The OverStitchTM Endoscopic Suturing System (Apollo Endosurgery, Inc. Austin, Texas) is an approved device designed to endoscopic placement of suture(s) and approximation of soft tissue. This system offers the assistant doctor the ability to restrict gastric pouch size by approximating tissue endoluminally through an incisionless (per-oral) approach. The use of this system has the potential to reduce the complications associated with the current surgical approach but still reaching the desired gastric restriction. The OverStitch has safely been used clinically for a great number of procedures that demanded an incisionless or minimally invasive approach, including endoluminal revisions for post-bypass gastric stoma and/or pouch dilatation, post-bypass fistulae repair, and oversewing of marginal ulcers.

Besides this suturing device, other endoscopic methods have already been used to reduce dilated stoma. Among them, ablation with argon plasma coagulation (APC) is one of the most important since this device is worldly available and presents an acceptable cost. Recent studies associate APC prior to endoscopic suture and initial evidence supports superiority of this association.

However, literature is still lacking of studies to support the use of APC associated with endoscopic suturing instead of APC alone. Therefore, the main focus of this study is to directly compare short and long-term effectiveness and safety of APC versus APC plus Endoscopic Full-thickness suture with OverStitch device in patients suffering from weight regain following RYGB.

Moreover, gut hormones regulation regarding bariatric and revisional procedures have been studied recently and evidence suggests that hormonal changes may be an important factor in weight loss. Three of the most important gut hormones regarding weight balance are ghrelin, GLP1 and peptide YY. Ghrelin is known as hunger hormone. It is produced by cells in gastric fundus. Glucagon-like Peptide 1 (GLP1) and Peptide YY (PYY) are both hormones that regulate satiety and are produced by L cells along distal intestine. Evidence in bariatric show that after long-term ghrelin levels diminish while GLP and PYY reach higher post-prandial peak. Regarding revisional endoscopic therapy, gut hormone changes have never been studied. That is also focus of this study as secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has stoma dilation defined as greater than 12mm, assessed with an esophagogastroduodenoscopy performed pre-operatively
2. Subject is ≥ 18 yrs. of age and ≤ 60 yrs. of age
3. Subject has a BMI of > 30
4. Subject has history of obesity for > 2 yrs
5. Subject has had no significant weight change (<5% of total body weight) in last 6 months
6. Subject must have failed standard obesity therapy (diet, exercise, behavior modification, and pharmacologic agents either alone or in combination), which will be assessed through an interview performed by a team member of the study at baseline
7. Subject is a reasonable candidate for general anesthesia
8. Subject agrees not to have any additional weight loss surgery or reconstructive surgery that may affect body weight (i.e. mammoplasty, liposuction, lipoplasty, etc) during the trial
9. Subject must be willing and able to participate in all aspects of the study and agree to comply with all study requirements for the duration of the study. This includes availability of reliable transportation and sufficient time to attend all follow-up visits.
10. Subject must be able to fully understand and be willing to sign the informed consent.

Exclusion Criteria:

1. Subject has had significant weight loss in the last 3 months, or between baseline and the study procedure
2. Mallampati (intubation) score greater than 3
3. Subject is observed during esophagogastroduodenoscopy to have heavily scarred, malignant or poor quality/friable tissue in areas of the stomach where sutures are to be placed
4. Subject has history of inflammatory disease of GI tract
5. Subject has a history of intestinal strictures or adhesions
6. Subject has renal and/or hepatic insufficiency
7. Subject has chronic pancreatic disease
8. Subject has history of/or signs and/or symptoms of gastro-duodenal ulcer disease and/or active peptic ulcer
9. Subject has significant esophageal disease including Zenker's diverticulum, grade 3-4 reflux esophagitis, stricture, Barrett's esophagus, esophageal cancer, esophageal diverticulum, dysphagia, achalasia, or symptoms of dysmotility
10. Subject has a history of any significant abdominal surgery
11. Subject has had previous bariatric, gastric or esophageal surgery; intestinal obstruction; portal gastropathy; gastrointestinal tumors; esophageal or gastric varices, or gastroparesis
12. Subject has a hiatal hernia > 2cm
13. Subject has chronic/acute upper GI bleeding conditions
14. Subject has severe coagulopathy (prothrombin time > 3 seconds over control or platelet count < 100,000) or is presently taking heparin, coumadin, warfarin, or other anticoagulants or other medications which impede coagulation or platelet aggregation, if they cannot be ceased for the procedure
15. Female subject is of childbearing age and not practicing effective birth control, is pregnant or is lactating
16. Subject has symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
17. Subject has cancer or life expectancy of < 2 yrs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Absolute Weight Loss | This outcome will be assessed at 12 months after the procedure
  Absolute Weight Loss will be assessed through subtraction of the pre-operative weight and the weight at follow-up, and will be measured in kilograms (kgs).
Excess Weight Loss | This outcome will be assessed at 12 months after the procedure
  Excess Weight Loss will be assessed through calculation of the percentage of the overweight lost after the procedure at follow-up. Excess Weight is defined as the weight over BMI of 25 for each patient. Excess Weight Loss will be expressed as percentage (%).
Abdominal Circumference Reduction | This outcome will be assessed at 12 months after the procedure
  Subtraction between baseline abdominal circumference and this measure at follow-up. This outcome will expressed in centimeters (cm).
BMI reduction | This outcome will be assessed at 12 months after the procedure.
  Subtraction between baseline BMI and this measure at follow-up. This outcome will expressed in kg/m2.
Diabetes improvement | This outcome will be assessed at baseline and 12 months after the procedure.
  This outcome will be assessed through a glucose tolerance test performed at baseline and another one performed at 1 year follow-up.

SECONDARY OUTCOMES:
Occurrence of Adverse Events | This outcome will be assessed continually after the procedure.
  Adverse events such as perforation, bleeding, pain, stenosis, vomiting, need of surgery.
Quality of Life Improvement | This outcome will be assessed at baseline and at 12 months.
  This outcome will be assessed with SF-36 questionnaire.
Eating Habits Evaluation | This outcome will be assessed at baseline and at 12 months.
  This outcome will evaluate if there is any change in eating habits with TFEQ-R21 questionnaire
Gut Hormones Response | This outcome will be assessed at baseline and at 12 months.
  This outcome will evaluate at fasting, 30, 60, 90 and 120 minutes post-prandial the hormonal variation regarding Ghrelin, GLP1 and PYY
Gastric (Pouch) Emptying | This outcome will be assessed at baseline and at 12 months.
  This outcome will evaluate retention rate through scintigraphy.
CT Volumetry of the Gastric Pouch | This outcome will be assessed at baseline and at 12 months.
  This outcome will evaluate volumetry of the pouch before and 12 months after procedure through tridimensional computed tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Vitor O Brunaldi, MD, Study Chair — University of Sao Paulo General Hospital; Eduardo G Hourneaux de Moura, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brunaldi VO, Farias GFA, de Rezende DT, Cairo-Nunes G, Riccioppo D, de Moura DTH, Santo MA, de Moura EGH. Argon plasma coagulation alone versus argon plasma coagulation plus full-thickness endoscopic suturing to treat weight regain after Roux-en-Y gastric bypass: a prospective randomized trial (with videos). Gastrointest Endosc. 2020 Jul;92(1):97-107.e5. doi: 10.1016/j.gie.2020.03.3757. Epub 2020 Mar 23. PMID 32217111